CLINICAL TRIAL: NCT00244777
Title: Introduction of New Hypo-osmolar ORS Into Routine Use in the Management of Diarrhoeal Disease: a Phase IV Clinical Surveillance.
Brief Title: Introduction of Hypo-osmolar ORS for Routine Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002-026
Record Dates: First submitted 2005-10-26; First posted 2005-10-27 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2005-10

CONDITIONS: Diarrhoea
Keywords: Seizure; Altered consciousness; Hyponatraemia; Diarrhoea; Hypo osmolar ORS
MeSH Terms: conditions — Diarrhea; Seizures; Hyponatremia

INTERVENTIONS:
Drug: Hypo-osmolar ORS

SUMMARY:
The World Health Organization has very recently recommended the routine use of a hypo-osmolar ORS in the management of diarrhoeal diseases. This recommendation is based on the better efficacy of the hypo-osmolar ORS over the standard WHO ORS demonstrated in controlled clinical trials. The recommendation, however, also expressed the need for "careful monitoring to better assess risk, if any, of symptomatic hyponatraemia". There thus is a need for phase IV trials before the new solution is introduced into routine clinical practice to assess the risk in relatively large number of patient populations. The proposed study will be carried out at two different settings- at the urban settings of the Dhaka Hospital (60000 patients) and at the rural settings of the Matlab Hospital (15000 patients) of ICDDR,B. The hypo-osmolar rice or glucose-based ORS will be introduced as standard management of patients with diarrhoea . The hypo-osmolar ORS will contain 75 mmol /L of sodium instead of 90 mmol/L. Surveillance will be carried out to detect adverse events focusing on the occurrence of seizures or undue lethargy during hospitalization. Each episode of seizure or undue lethargy would be evaluated to determine if they are associated with abnormal levels of serum sodium or glucose, or fever. It has been estimated that about 3% (1,800) of patients initially admitted to the Short Stay Ward of the Dhaka Hospital, and 340 patients at the Matlab Hospital might require admission to the longer stay inpatient wards due to seizure or altered consciousness. Such patients would be thoroughly assessed including determination of their serum sodium and glucose, two common causes of seizures/altered consciousness, to determine if and to what extent they could be attributed to hyponatraemia.The results from this study would be used in planning and implementing the routine use of the new formulation of ORS at all Government, NGO and private health care facilities that treat diarrhoeal patients, in Bangladesh and in other countries.

DETAILED DESCRIPTION:
Study site: The Dhaka and the Matlab Hospitals of ICDDR, B: Centre for Health and Population Research.

Duration: Total duration of 15 months that include data collection over a full year to capture seasonal variations in the aetiology of diarrhoea.

Sample size: Based on the yearly patient visits it is estimated that 60,000 patients would be studied at the Dhaka Hospital and 15,000 patients at the Matlab Hospital.

Inclusion criteria

All patients attending the Dhaka and Matlab hospitals who will be admitted to the Short Stay Ward with uncomplicated watery diarrhoea would be eligible for this study.

Exclusion criteria

Patients with complications, and those with severe illness that require special care or multiple interventions would be excluded.

Procedures

Infants 6 month of age or younger would receive the glucose-based (75 mmol/L) ORS ( Na: 75, Cl: 65, K: 20, citrate:10, glucose: 75, and osmolarity: 245 mOsm/L), and those older than 6 months would receive the rice-based ORS (40 g/L of rice powder); both will contain 75 mmol/L of sodium, 65 mmol/L of chloride, 20 mmol/L of potassium, and 10 mmol/L of citrate with an in vitro osmolarity of 170 mOsm/L. This is in line with the Centre's policy of not adding starch for management of infants 6 months of age or younger.

Surveillance and case management

Dhaka Hospital: From our experience about 3% patients (1,800 patients/year) initially admitted to the Short Stay Ward are subsequently admitted to the Longer Stay Wards due to development of symptoms like seizure, lethargy or altered consciousness. Patients admitted to the Short Stay Ward who receive ORS solution for 8 hours or more, and subsequently admitted to inpatient ward for the above symptoms will be evaluated to determine if they are due to hyponatraemia. Similarly, 3% of the patients attending the Matlab Hospital (340 patients/year) might develop these symptoms and will be evaluated if their symptoms are due to hyponatraemia.

All clinical and laboratory data of these patients will be maintained during the study.

Assessment and management of patients Hospitals current protocol for assessment of the cause of lethargy and seizures such as estimation of plasma glucose, serum electrolytes, fever, and study of the cerebrospinal fluids where clinically indicated would be employed for diagnosing the aetiology of the symptoms.

Protocol for management of seizure

Although rare, the development of seizures during the rehydration therapy for acute watery diarrhoea would be considered as a serious adverse event. Patients developing such symptoms would be assed to determine if they could be attributed to hyponatraemia. The same protocol for management of seizure would be used at both of the study sites, which would be as follows:

Procedures:

* All patients developing significant lethargy and seizure while on ORS would be immediately admitted to the special care unit.
* An intravenous line will be opened for medication.
* Blood glucose will be measured immediately from finger blood sample using bedside glucose monitoring machine, and blood sample would be obtained for estimation of serum electrolytes, calcium, and magnesium at the clinical laboratories of the Centre.
* Hypoglycaemic (<2.2 mmol/L) patients would be immediately given intravenous glucose (25% glucose; 2 ml/kg), which would be followed by oral (or through nasogastric tube of patients who are unable to drink) administration of 10% glucose in a dose of xxxxx
* Diazepam (0.3 mg/Kg) would be administered to patients who are not hypoglycaemia, and also to patients who are hypoglycaemic but do not respond to initial glucose infusion.
* If seizure persists, the same dose of intravenous diazepam would be repeated for the second time, and injectable phenobarbitone would also be administered (15-20 mg/kg loading dose, followed by 2.5 mg/Kg every 12 hours as the maintenance dose).
* After control of seizure, a lumber tap will be done to rule out meningitis if clinically indicated (i.e. patients suspected to have meningitis).
* A sample of blood will also be sent for culture to exclude septicaemia
* X-Ray chest will be done to exclude pneumonia if clinically indicated (following WHO guidelines)
* Patients with a serum sodium of ≤120 mmol/L will be treated with 3% NaCl in a dose of 1 ml/Kg.hour for the next 4 hours (i.e. total of 12 ml/Kg over the 4-hour period), along with restriction of plain water.
* Hypernatraemic patients (serum sodium >150 mmol/L) would be treated with the same ORS but with provision for water ad lib.
* Patients suspected for extra intestinal infection including sepsis will be treated with Inj. Ampicillin and Inj. Gentamicin (infants aged 3 months or younger) or Inj. Ceftriaxone and Gentamicin (patients aged more than 3 months) for 7 days.

ELIGIBILITY:
Inclusion Criteria:

All age group Either sex Acute watery diarrhoea

Exclusion Criteria:

Diarrhoea with complication and other severe illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75000
Dates: Start 2002-12; Primary Completion 2004-02 (Actual); Study Completion 2004-02

PRIMARY OUTCOMES:
Incidence of symptomatic ( seizure/altered conciousness)hyponatremia(serum sodium < 130 m.mol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Nur H Alam, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh